CLINICAL TRIAL: NCT00506974
Title: Enhancing Slow Wave Sleep With Sodium Oxybate to Reduce the Behavioral and Physiological Impact of Sleep Loss
Brief Title: Enhancing Slow Wave Sleep With Sodium Oxybate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Dr. Paula Schweitzer, St. Luke's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2007.002
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Sleep
Keywords: sleep; normal sleepers
MeSH Terms: interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sodium oxybate — 3.5 g of sodium oxybate or placebo on two of the five overnights.
  Other Names: xyrem

SUMMARY:
The purpose of this study is to determine if there the impact of sleep deprivation upon sleepiness, attention, memory, and mood is reduced by pharmacologically enhancing slow wave sleep (SWS) with sodium oxybate.

DETAILED DESCRIPTION:
SWS has been hypothesized to be a time of relatively high neural recuperation from wakefulness. That hypothesis has been prompted by a number of observations, including: 1) enhanced SWS following sleep deprivation in proportion to the duration of prior wakefulness, 2) reduced amounts of SWS during nocturnal sleep following afternoon/evening naps, 3) a gradual decline in SWS across a night of sleep, and 4) increased SWS following nights of fragmented sleep. Within the two-process model of sleep regulation, heightened SWS has been viewed as reflecting Process S, the homeostatic component. Many authors have proposed that increased SWS represents ongoing cortical recovery from prior wakefulness activities and is a time of relatively heightened neurophysiologic restoration or recuperation. In a prior study which we conducted (Walsh et al., 1994) there was a suggestion, from post hoc analyses, that SWS may prevent adverse effects of sleep loss. Additionally, we recently published the results of an investigation of pharmacologically-enhanced SWS (with tiagabine) during sleep restriction which demonstrated preserved neurobehavioral performance despite sleep restriction (Walsh et al, 2006). In the proposed research we will examine whether pharmacological enhancement of SWS with sodium oxybate reduces the impact of sleep deprivation upon sleepiness, attention, performance, mood, and autonomic nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

1. males and females, ages 18-50 inclusive
2. use of adequate contraceptive procedures throughout the study for females.

Exclusion Criteria:

1. pregnancy or lactating
2. prior use of or allergy to sodium oxybate
3. participation in a clinical research trial within the past 30 days
4. blood donation within the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
MSLT | throughout the study
PVT | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: James K Walsh, Ph.D., Principal Investigator — Sleep Medicine and Research Center at St. Luke's Hospital
Locations (1):
- Sleep Medicine and Research Center at St. Luke's Hospital, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Walsh JK, Hartman PG, Schweitzer PK. Slow-wave sleep deprivation and waking function. J Sleep Res. 1994 Mar;3(1):16-25. doi: 10.1111/j.1365-2869.1994.tb00099.x. PMID 10607104
- [Background] Walsh JK, Randazzo AC, Stone K, Eisenstein R, Feren SD, Kajy S, Dickey P, Roehrs T, Roth T, Schweitzer PK. Tiagabine is associated with sustained attention during sleep restriction: evidence for the value of slow-wave sleep enhancement? Sleep. 2006 Apr;29(4):433-43. PMID 16676776